CLINICAL TRIAL: NCT03752359
Title: Effect of Whey Protein Supplementation Combined With Resistance Training on Body Composition, Muscular Strength, Functional Capacity, and Plasma-metabolism Biomarkers in Older Women With Sarcopenic Obesity
Brief Title: Whey Protein Supplementation and Resistance Training in Older Women With Sarcopenic Obesity.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Coordination for the Improvement of Higher Education Personnel (Other)
Responsible Party: Principal Investigator, Hellen Clair Garcêz Nabuco, Principal Investigator, Universidade Estadual de Londrina
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: UEL1700756-1/2018
Record Dates: First submitted 2018-11-16; First posted 2018-11-26 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Body Weight; Healthy
Keywords: sarcopenia; obesity; protein intake; IL-6; lean tissue
MeSH Terms: conditions — Body Weight; Sarcopenia; Obesity | interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- whey protein group (Experimental): Participants received a dose of 35 grams of whey protein after resistance training (RT). Participants were personally supervised by physical education professionals with substantial RT experience. The sessions were performed 3 times per week on Mondays, Wednesdays, and Fridays, with 3 sets of 08-12 repetition maximums. The RT program was a whole-body program with eight exercises, including: chest press, seated row, triceps push-down, preacher curl, horizontal leg press, knee extension, leg curl and seated calf raise. Participants were afforded a 1 to 2 min rest interval between sets and 2 to 3 min between each exercise. The training load was consistent with the prescribed number of repetitions for the three sets of each exercise.
  Interventions: Dietary Supplement: whey protein
- placebo group (Placebo Comparator): Participants received a dose of 35 grams of maltodextrin after resistance training (RT). Participants were personally supervised by physical education professionals with substantial RT experience. The sessions were performed 3 times per week on Mondays, Wednesdays, and Fridays, with 3 sets of 08-12 repetition maximums. The RT program was a whole-body program with eight exercises, including: chest press, seated row, triceps push-down, preacher curl, horizontal leg press, knee extension, leg curl and seated calf raise. Participants were afforded a 1 to 2 min rest interval between sets and 2 to 3 min between each exercise. The training load was consistent with the prescribed number of repetitions for the three sets of each exercise.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: whey protein — This two-arm randomized, double-blind, placebo-controlled design was carried out over a period of 16 weeks. At the beginning and end of the experiment, two weeks were allocated for evaluations consisting of anthropometric (weeks 2 and 16), body composition (weeks 2 and 16), one repetition maximum tests (weeks 1 and 15), functional capacity tests (weeks 1 and 15), blood samples (weeks 2 and 16) and dietary intake measurements (weeks 1 and 15). The anthropometric, body composition, blood samples and dietary intake measurements were carried out in a temperature-controlled room (22-24 °C), and the RT sessions were conducted at the university training facility.
  Arms: whey protein group
Dietary Supplement: placebo — This two-arm randomized, double-blind, placebo-controlled design was carried out over a period of 16 weeks. At the beginning and end of the experiment, two weeks were allocated for evaluations consisting of anthropometric (weeks 2 and 16), body composition (weeks 2 and 16), one repetition maximum tests (weeks 1 and 15), functional capacity tests (weeks 1 and 15), blood samples (weeks 2 and 16) and dietary intake measurements (weeks 1 and 15). The anthropometric, body composition, blood samples and dietary intake measurements were carried out in a temperature-controlled room (22-24 °C), and the RT sessions were conducted at the university training facility.
  Arms: placebo group

SUMMARY:
The main purpose of the present study was to investigate the effects of whey protein following resistance training on body composition, muscular strength, functional capacity, and plasma-metabolism biomarkers in older women with sarcopenic obesity.

DETAILED DESCRIPTION:
This two-arm randomized, double-blind, placebo-controlled design was carried out over a period of 16 weeks. At the beginning and end of the experiment, two weeks were allocated for evaluations consisting of anthropometric (weeks 2 and 16), body composition (weeks 2 and 16), one repetition maximum tests (weeks 1 and 15), functional capacity tests (weeks 1 and 15), blood samples (weeks 2 and 16) and dietary intake measurements (weeks 1 and 15). The anthropometric, body composition, blood samples and dietary intake measurements were carried out in a temperature-controlled room (22-24 °C), and the RT sessions were conducted at the university training facility.

Recruitment was carried out through newspapers, radio advertising, and home delivery of leaflets in the central area and residential neighborhoods. All participants completed health history and physical activity questionnaires and were included in the study if they met the following inclusion criteria: 60 years old or more, physically independent, free from cardiac or orthopedic dysfunction that would prevent them from performing the prescribed exercise or exercise testing associated with the study, not receiving hormonal replacement therapy, and completed a previous 8-week RT program. In this study, only women with SO were included. SO was defined as a body fat mass ≥ 35%(29) combined with appendicular lean soft tissue (ALST) less than <15.02 kg(30), assessed by dual x-ray energy absorptiometry (DXA). Participants underwent a diagnostic graded exercise stress test with a 12-lead electrocardiogram reviewed by a cardiologist and were released with no restrictions for participation in this investigation.

A blinded researcher was responsible for generating random numbers for participant allocation. Both groups were submitted to the same RT program and all participants completed the experiment. Written informed consent was obtained from all participants after a detailed description of investigation procedures was provided. This investigation was conducted according to the Declaration of Helsinki and was approved by the local University Ethics Committee The Shapiro Wilk test was used to test data distribution. Data are presented as means, standard deviation, and z-score. The student's independent t-test and chi-square test were used to compare groups regarding the general characteristics and clinical/medical history (categorical variables). Two-way analysis of variance (ANOVA) for repeated measures was used to assess between group comparisons. The effect size (ES) was calculated to verify the magnitude of the differences by Cohen's d, where an ES of 0.20-0.49 was considered as small, 0.50-0.79 as moderate, and ≥ 0.80 as large(41). The Z-score of the percentage changes (from pre- to post-training) of the raw data for each parameter was calculated, as well as a total Z-score, derived from all the components. To verify the differences between groups in total Z-scores, an independent T test was also applied. For all statistical analyses, significance was accepted at P < 0.05. The data were analyzed using SPSS software version 20.0 (SPSS, Inc., Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

60 years old or more, physically independent, free from cardiac or orthopedic dysfunction that would prevent them from performing the prescribed exercise or exercise testing associated with the study, not receiving hormonal replacement therapy, and completed a previous 8-week RT program. In this study, only women with SO were included. SO was defined as a body fat mass ≥ 35% combined with appendicular lean soft tissue (ALST) less than <15.02 kg, assessed by dual x-ray energy absorptiometry (DXA). Participants underwent a diagnostic graded exercise stress test with a 12-lead electrocardiogram reviewed by a cardiologist and were released with no restrictions for participation in this investigation.

Exclusion Criteria:

All subjects not participating in 85% of the total sessions of training or withdraw

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2017-03-17 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Change in body composition | baseline and after 12 weeks
  Whole-body dual-energy X-ray absorptiometry (DXA) (Lunar Prodigy) was used to assess lean mass and fat mass and its segments. The total skeletal muscle mass (SMM) was estimated by the predictive equation proposed by Kim et al. (Kim et al., 2004). The results are presented in kg.
Change in Muscular strength | baseline and after 12 weeks
  Maximal dynamic strength was evaluated using the 1RM test assessed on chest press, knee extension, and preacher curl exercises performed in this exact order. Testing for each exercise was preceded by a warm-up set (6-10 repetitions), with approximately 50% of the estimated load used in the first attempt of the 1RM. This warm-up was also used to familiarize the subjects with the testing equipment and lifting technique. The testing procedure was initiated 2 minutes after the warm-up. The subjects were instructed to try to accomplish two repetitions with the imposed load in three attempts in both exercises. The rest period was 3 to 5 min between each attempt, and 5 min between exercises. The 1RM was recorded as the last resistance lifted in which the subject was able to complete only one single maximal execution

SECONDARY OUTCOMES:
Change in inflammatory markers | baseline and after 12 weeks
  Tumor Necrosis Factor -α (TNF-α) and Interleukin-6 (IL-6) were determined by enzyme-linked immunosorbent assay (ELISA), according to the specifications of the manufacturer and performed in a microplate reader Perkin Elmer, model EnSpire (USA). All samples were determined in duplicate to guarantee the precision of the results. The results are presented in picograms per milliliter (pg/ml).
Change in C-reactive protein (CRP) | baseline and after 12 weeks
  Measurements of serum levels of high-sensitivity CRP were carried out using a biochemical auto-analyzer system (Dimension Max - Siemens Dade Behring) according to established methods in the literature consistent with the manufacturer's recommendations. The results are presented in milligrams per decilitre (mg/dL).
Change in oxidative stress | baseline and after 12 weeks
  For measurements, advanced oxidation protein products (AOPP) were determined in the plasma using a semiautomatic method. AOPP concentrations were expressed as micromoles per liter (μmol/L). Total plasma antioxidant capacity (TRAP) was determined by the chemiluminescence method for the induction time of 2.2 azo-bis (2-amidinopropane) and calibrated with Trolox analogue of vitamin E. TRAP values were expressed in μmol of Trolox.
Change in Total cholesterol | baseline and after 12 weeks
  Measurements of serum levels of total cholesterol were determined using a biochemical auto-analyzer system (Dimension Max - Siemens Dade Behring) according to established methods in the literature consistent with the manufacturer's recommendations.
Change in high-density lipoprotein (HDL-C) | baseline and after 12 weeks
  Measurements of serum levels of high-density lipoprotein were determined using a biochemical auto-analyzer system (Dimension Max - Siemens Dade Behring) according to established methods in the literature consistent with the manufacturer's recommendations.
Change in triglycerides | baseline and after 12 weeks
  Measurements of serum levels of triglycerides were determined using a biochemical auto-analyzer system (Dimension Max - Siemens Dade Behring) according to established methods in the literature consistent with the manufacturer's recommendations.
Change in low-density lipoprotein | baseline and after 12 weeks
  For the determination of LDL-c was used the Friedewald equation: LDL-c=TC - (HDL-c + TG / 5).
Change in glucose | baseline and after 12 weeks
  Measurements of serum levels of glucose (GLU) were determined using a biochemical auto-analyzer system (Dimension Max - Siemens Dade Behring).
Change in insulin | baseline and after 12 weeks
  Insulin was determined by the chemiluminescence method (LIASON equipment)
Change in HOMA-IR | baseline and after 12 weeks
  The Homeostasis Assessment Model (HOMA-IR) was calculated by the formula: Insulin fasting (μUI / mL) x Glucose fasting (mmol / L) / 22.5.
Change in blood pressure | baseline and after 12 weeks
  Resting BP assessment was performed using automatic, oscillometric equipment (Omron - 7113). Participants attended the laboratory on three different days and, during each visit, remained seated at rest for 10 min with the cuff of the equipment in place on the right arm. Subsequently, several BP measurements were performed at one-minute intervals in order to obtain three consecutive measurements where the difference in systolic BP (SBP) and diastolic BP (DBP) readings differed by no more than 4 mmHg. The average of the three measurements for each day was averaged across the three visits.
Change in body mass | baseline and after 12 weeks
  Body mass was measured to the nearest 0.1 kg using a calibrated electronic scale, with subjects wearing light workout clothing and no shoes.
Change in height | baseline and after 12 weeks
  Height was measured using a stadiometer to the nearest 0.1 cm while subjects were standing without shoes.
Change in body mass index | baseline and after 12 weeks
  Body mass index was calculated as the body mass in kilograms divided by the square of the height in meters.
Change in waist circumference | baseline and after 12 weeks
  We also collected data on waist circumference (WC), using a flexible and inelastic tape measure. WC was obtained at the midpoint between the last rib and the iliac crest at the time of expiration. Two measurements were used to measure each circumference. In situations in which the difference between the measurements was greater than 0.5 cm a third measurement was performed, with the value of the median being adopted as reference. All measurements were performed by the same evaluator.
Change in hip circumference | baseline and after 12 weeks
  We also collected data on hip circumference, using a flexible and inelastic tape measure. HC was measured in the region of greater perimeter between the waist and the thigh. Two measurements were used to measure each circumference. In situations in which the difference between the measurements was greater than 0.5 cm a third measurement was performed, with the value of the median being adopted as reference. All measurements were performed by the same evaluator.
Dietary intake | baseline and after 12 weeks
  Food consumption were assessed by the 24-hour dietary recall method applied on two non-consecutive days of the week, with the aid of a photographic record taken during an interview. The homemade measurements of the nutritional values of food and supplementation were converted into grams and milliliters by the online software Virtual Nutri Plus for diet analysis. Some foods were not found in the program database and therefore items were added from food tables.

CONTACTS AND LOCATIONS:
Overall Officials: Edilson Cyrino, PhD., Study Director — Universidade Estadual de Londrina
Locations (1):
- Hellen Clair Garcez Nabuco, Cuiabá, Mount, Brazil

REFERENCES:
- [Background] American College of Sports Medicine. American College of Sports Medicine position stand. Progression models in resistance training for healthy adults. Med Sci Sports Exerc. 2009 Mar;41(3):687-708. doi: 10.1249/MSS.0b013e3181915670. PMID 19204579
- [Background] Kim J, Heshka S, Gallagher D, Kotler DP, Mayer L, Albu J, Shen W, Freda PU, Heymsfield SB. Intermuscular adipose tissue-free skeletal muscle mass: estimation by dual-energy X-ray absorptiometry in adults. J Appl Physiol (1985). 2004 Aug;97(2):655-60. doi: 10.1152/japplphysiol.00260.2004. Epub 2004 Apr 16. PMID 15090482
- [Background] Sardinha LB, Lohman TG, Teixeira PJ, Guedes DP, Going SB. Comparison of air displacement plethysmography with dual-energy X-ray absorptiometry and 3 field methods for estimating body composition in middle-aged men. Am J Clin Nutr. 1998 Oct;68(4):786-93. doi: 10.1093/ajcn/68.4.786. PMID 9771855
- [Derived] Nabuco HCG, Tomeleri CM, Fernandes RR, Sugihara Junior P, Cavalcante EF, Cunha PM, Antunes M, Nunes JP, Venturini D, Barbosa DS, Burini RC, Silva AM, Sardinha LB, Cyrino ES. Effect of whey protein supplementation combined with resistance training on body composition, muscular strength, functional capacity, and plasma-metabolism biomarkers in older women with sarcopenic obesity: A randomized, double-blind, placebo-controlled trial. Clin Nutr ESPEN. 2019 Aug;32:88-95. doi: 10.1016/j.clnesp.2019.04.007. Epub 2019 May 13. PMID 31221297